CLINICAL TRIAL: NCT04163276
Title: Creation of a Database of PET Digital Brain Exams, Adapted to a Population Aged 50 Years and Over, to Help in the Interpretation of Fluoro Desoxy Glucose (FDG) Labelled With Fluor 18 (18F-FDG) PET/CT (Computer Tomography) Exam
Brief Title: Database of Positon Emission Tomography (PET) Digital Brain Exams, in 50th Age of Patients
Acronym: BASITEP
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: GIE NANCYCLOTEP (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI238
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Neurodegenerative Diseases
Keywords: neurodegenerative disease; digital brain PET exam; database
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: 20 patients without anomaly of brain metabolism
  Interventions: Diagnostic Test: 18F FDG PET exam
- Group 2: 20 patients with Alzheimer's disease
  Interventions: Diagnostic Test: 18F FDG PET exam

INTERVENTIONS:
Diagnostic Test: 18F FDG PET exam — All patients have received 18F-FDG PET/CT in nuclear medicine

SUMMARY:
This study evaluate the interest to create a new database of PET digital brain exams in population of 50 years and over of patients. Half of patients with no abnormal brain metabolism while the other half patients with Alzheimer's disease.

DETAILED DESCRIPTION:
The 18F-FDG cerebral PET can be performed for the detection of neurodegenerative diseases found hypometabolism in the areas concerned (Alzheimer's disease, fronto-temporal dementia, dementia Lewy body etc). The diagnosis is given by the clinician with a visual analysis of the data. Technical aids are now recommended (European recommendations) to complete the diagnosis with a quantitative analysis of different brain regions to a healthy brain base, to guide the diagnosis, in addition to visual analysis.

The emergence of a new technology has allowed the transition from analog PET / CT to digital PET / CT improving spatial resolution and image contrast. Unlike analog PET / CT that uses photomultipliers to detect light, digital PET / CT uses the digital photon counting technique to directly convert light into a digital signal and each crystal is connected to a single detector.

Different software, used in clinical routine, gives access to a quantified analysis of different areas of the brain. However, these programs have been made with healthy subjects of reduced strength (for example, the Neuro Q ® software database is based on 29 healthy patients), with no specific age and thanks to analog PET / CT ( old generation). There is therefore a low specificity in terms of detection of degenerative pathologies, this being explained by a decrease in cerebral metabolism with age 9, mainly at the level of the anterior areas 10 (frontal lobe, temporopolar areas, insular areas, cortex anterior cingulate).

ELIGIBILITY:
Inclusion Criteria:

* Having performed a 18F-FDG cerebral PET/CT exam as part of an Alzheimer's assessment at the Nuclear Medicine department of NANCY, sent by the Geriatric Department
* Patient who has received complete information on the organization of the research and who has not objected to the exploitation of this data
* Patient affiliated to a social security

Exclusion Criteria:

* patient who has received complete information on the organization of the research and who has objected to the exploitation of this data
* For patients with no abnormality in 18F-FDG PET, Mini Mental State Examination (MMSE) <25 or clinically diagnosed neurodegenerative pathology
* For patients with typical hypometabolism of 18F-FDG PET/CT, biology of cerebrospinal fluid not in favor of Alzheimer's disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population will be enrolled thank to a listing of patient available in nuclear médicine unit. This listing cntain patient who performed a 18F-FDG brain TEP in nuclear médicine unit between 2010 and 2019.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-01-02 (Actual); Primary Completion 2020-06-06 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
data base analysis | 1 hour
  Comparison of Z-scores from PET/CT of the quantitative analysis of patients without abnormality of the brain metabolism and of typical Alzheimer patients (brain metabolism of the regions involved in Alzheimer's disease), calculated with 2 databases:
  * An analogue database consisting of 18F-FDG PET/CT without brain metabolism abnormalities in patients aged 50 and over;
  * A digital database, consisting of 18F-FDG PET/CT without brain metabolism abnormalities in patients aged 50 and over

CONTACTS AND LOCATIONS:
Overall Officials: Verger Antoine, PhD, Study Chair — Central Hospital, Nancy, France
Locations (1):
- University hospital of Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No